CLINICAL TRIAL: NCT02060175
Title: Comparison of the 3-month Strut Coverage After Coronary Stenting by Optical Coherence Tomography; Cilotax and DESyne
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of the problem with Cilotax stent permission
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0076
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Patients in the Treatment of Subjects With All-comer Who Are to Undergo PCI
Keywords: Optical coherence tomography, Drug-eluting stent, Strut coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 CILOTAX arm (Experimental): Cilotax drug-eluting stents implantation
  Interventions: Device: Cilotax drug-eluting stents implantation
- 2 DESyne arm (Active Comparator): DESyne drug-eluting stents implantation
  Interventions: Device: DESyne drug-eluting stents implantation

INTERVENTIONS:
Device: Cilotax drug-eluting stents implantation
  Arms: 1 CILOTAX arm
Device: DESyne drug-eluting stents implantation
  Arms: 2 DESyne arm

SUMMARY:
We will compare the stent coverage at 3 months by optical coherence tomography (OCT) between the Cilotax and DESyne drug-eluting stents (DES). The extent of the strut uncoverage has not been evaluated yet for both the Cilotax and DESyne and we first sought to decide the reference intervals using 40 samples (total 44 patients for each group considering 10% drop-out rate) as the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 20 years old
* Patients in the treatment of subjects with all-comer who are to undergo PCI

Exclusion Criteria:

* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Stent coverage | up to 3 months after stent implantation
  The percentage of stent uncoverage measured by OCT